CLINICAL TRIAL: NCT04461847
Title: A Randomized Controlled Trial of Endoscopic Subcutaneous Mastectomy Versus Open Mastectomy in Early Breast Cancer Patients
Brief Title: ESM Versus OM ：A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigator, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFH-BC
Record Dates: First submitted 2020-04-07; First posted 2020-07-08 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Endoscopic Subcutaneous Mastectomy
MeSH Terms: interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients underwent ESM (Experimental)
  Interventions: Procedure: endoscopic subcutaneous mastectomy
- patients underwent SM (Active Comparator)
  Interventions: Procedure: subcutaneous mastectomy

INTERVENTIONS:
Procedure: subcutaneous mastectomy — Operating subcutaneous mastectomy
  Arms: patients underwent SM
Procedure: endoscopic subcutaneous mastectomy — Operating endoscopic subcutaneous mastectomy
  Arms: patients underwent ESM

SUMMARY:
The consideration of quality of life issues has led to the development of alternative surgeries for breast cancer patients, particularly in the case of localized disease. Nipple-sparing subcutaneous mastectomy (SM), for example, was designed to preserve the nipple-areola complex which facilitates breast reconstruction. However, SM still leaves behind a conspicuous scar.There have already been some observation study show that endoscopic subcutaneous mastectomy(ESM) can improve the cosmesis outcomes and at the same time as safe as the traditional SM.However there is no RCT in this field.That is why the investigators design this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stages I or II ductal carcinoma
2. The distance from the tumor to the edge of the papilla is more than 3cm, the tumor volume is less than 3cm, the axillary lymph nodes have no obvious fusion and no adhesion with the axillary vein and brachial plexus
3. Age from 18~70
4. ECOG scores 0~2
5. Normal function of liver, kidney and bone marrow

Exclusion Criteria:

1. Through physical examination and MRI, it was confirmed that the tumor did not invade the skin, but was confined to the gland and did not invade the surface of the gland.
2. There are serious medical diseases
3. Pregnant or lactating women women of childbearing age -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
local recurrence rate | 12 months after operation
  Definition and diagnostic criteria of local recurrence: physical examination or imaging examination found lesions in the same side of breast, chest wall or skin and surgical scars, and confirmed by histology as breast cancer of the same tissue type; 12 months after operation, the evaluation was carried out.

SECONDARY OUTCOMES:
Distant metastasis | 12 months after operation
  Definition and diagnosis criteria of distant metastasis: the lesions appeared in the distant organs other than breast and surrounding tissues, such as bone, lung, liver, brain, etc., and were diagnosed as breast cancer metastasis by imaging or histology; the evaluation was carried out 12 months after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang ZH, Ding G, Wu S, Song JN, Ge ZC, Zhang H, Yuan Z, Gao YG, Gang TR, Zhang Z, Qu X. Oncological outcome of single-port insufflation endoscopic nipple-sparing mastectomy versus open mastectomy in early breast cancer patients: a study protocol for a randomised controlled trial. BMJ Open. 2022 May 2;12(5):e047866. doi: 10.1136/bmjopen-2020-047866. PMID 35501091